CLINICAL TRIAL: NCT07368400
Title: Development and Investigation of the Effectiveness of a Gamified Mobile Physical Therapy Exercise Application for Children With Duchenne Muscular Dystrophy: A 6-Month Follow-Up Single-Blind Randomized Controlled Trial
Brief Title: DMD and Gamified Physiotherapy
Acronym: Gamified DMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başak Çağla Arslan (Other Government)
Collaborators: Hacettepe University (Other); Lokman Hekim University (Other Government); Bezmialem Vakif University (Other)
Responsible Party: Sponsor-Investigator, Başak Çağla Arslan, Lecturer, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 125S143; 125S143 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: dmd; exercise; gamification
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are randomly allocated to either an intervention group or a control group. The intervention group receives a gamified mobile physiotherapy exercise program in addition to center-based physiotherapy, while the control group receives the same center-based physiotherapy plus standard home exercise instructions. Since the effects of the intervention are expected to be unidirectional and may not be reversible in a short duration, a parallel model was chosen over a crossover design. The groups are followed simultaneously and do not cross over during the study. The model allows comparison of short-term treatment effects and longer-term adherence outcomes.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation to reduce assessment bias. Participants, caregivers, and treating clinicians were not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Mobile Physiotherapy + Center-Based Physiotherapy (Experimental): Participants assigned to the intervention arm will receive center-based physiotherapy three times per week for 8 weeks (45-minute sessions), in combination with a gamified mobile physiotherapy exercise application to be performed at home. The mobile component includes personalised exercise tasks, real-time feedback, and progression-based digital features to support home exercise completion. Participants will be instructed to use the application in accordance with a structured schedule provided by the clinical team.
  Interventions: Behavioral: Gamified Mobile Physiotherapy Exercise Application
- Standard Home Exercise + Center-Based Physiotherapy (Active Comparator): Participants assigned to the control arm will receive center-based physiotherapy three times per week for 8 weeks (45-minute sessions), in combination with standard home exercise instructions provided by the clinical team. Home exercises are prescribed according to conventional physiotherapy protocols for Duchenne muscular dystrophy and are to be performed without digital support.
  Interventions: Behavioral: Standard Home Exercise Instructions

INTERVENTIONS:
Behavioral: Gamified Mobile Physiotherapy Exercise Application — A mobile gamified exercise program designed for children with Duchenne muscular dystrophy. The program includes personalised exercise tasks, progression-based game features, and feedback to support home-based physiotherapy participation.
  Other Names: Center-Based Physiotherapy (Behavioral)
  Arms: Gamified Mobile Physiotherapy + Center-Based Physiotherapy
Behavioral: Standard Home Exercise Instructions — Conventional physiotherapy home exercise instructions provided as written and verbal guidance without digital or gamified components. Exercises are aligned with standard clinical practice for Duchenne muscular dystrophy.
  Arms: Standard Home Exercise + Center-Based Physiotherapy

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is a progressive neuromuscular disease that limits children's physical function, mobility, and participation in daily life. Regular physiotherapy and exercise are essential to slow functional decline; however, many children experience difficulties maintaining motivation and adherence to long-term exercise programs. Low adherence leads to reduced treatment benefit and faster loss of motor abilities.

This study aims to investigate whether a gamified mobile physiotherapy exercise program can improve participation, motivation, and physical outcomes in children with DMD. The mobile program includes personalized exercises designed by physiotherapists and occupational therapists, combined with game-based elements such as rewards, levels, feedback, and virtual achievements to enhance engagement. The program is delivered in addition to face-to-face physiotherapy.

A total of 46 boys aged 6-12 years with a confirmed diagnosis of DMD will be recruited and randomly assigned to either an intervention group or a control group. Both groups will attend an 8-week center-based physiotherapy program. The intervention group will additionally use the gamified mobile exercise application at home, while the control group will receive a standard home exercise program. Participants will be evaluated before treatment, after 8 weeks, and at 6-month follow-up.

The primary outcomes include physical function, endurance, and mobility. Secondary outcomes include psychosocial well-being, motivation, and therapy participation. The study intends to determine whether gamification-based telerehabilitation can increase adherence, preserve physical abilities, and support participation in children with DMD. If effective, this approach may offer a practical and accessible tool to support long-term rehabilitation needs in this population.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a progressive neuromuscular disorder that leads to loss of muscle strength, functional decline, reduced mobility, and limitations in participation. Early and ongoing physiotherapy is essential to slow functional deterioration, maintain mobility, and support participation in daily-life activities. Despite its importance, adherence to long-term exercise programs is frequently low among children with DMD due to fatigue, monotony, lack of feedback, limited motivation, and challenges related to time management and caregiver burden.

Gamification has emerged as a promising method to sustain motivation and engagement by integrating game-based elements such as challenges, levels, rewards, feedback, and achievement-based progression into non-game health contexts. Digital and mobile health solutions also provide an opportunity to deliver personalised and home-based rehabilitation, support remote follow-up, and increase continuity of care. However, evidence for gamified telerehabilitation specifically designed for DMD is limited, and most existing telerehabilitation programs lack systematic motivational components or long-term follow-up data.

This study evaluates a gamified mobile physiotherapy exercise program developed for children with DMD to increase motivation, participation, and adherence to home-based rehabilitation. The program includes personalised exercise tasks designed by physiotherapists and occupational therapists, and integrates gamification mechanisms to reinforce engagement. The intervention is delivered alongside an 8-week center-based physiotherapy program and followed for an additional 6 months to assess long-term adherence and carry-over effects.

A total of 46 boys aged 6-12 years with a confirmed diagnosis of DMD will be recruited and randomly assigned to an intervention group or a control group. Both groups receive an identical center-based physiotherapy program, whereas the intervention group additionally uses the mobile application at home. The control group receives standard home-exercise instructions. Assessments occur at baseline, post-intervention, and at a 6-month follow-up.

Primary outcomes focus on physical function, mobility, and endurance. Secondary outcomes include psychosocial well-being, motivation, and therapy participation. This study aims to determine whether a gamified telerehabilitation approach can enhance adherence, help preserve physical function, and support participation in children with DMD. If effective, this digital model may offer an accessible, motivating, and scalable strategy for long-term rehabilitation in pediatric neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male child aged 6 to 12 years with a confirmed diagnosis of Duchenne muscular dystrophy (DMD) based on specialist evaluation and genetic testing.
* Vignos lower extremity classification stage 1 or 2.
* Brooke upper extremity functional classification at least stage 5.
* Score of 27 or higher on the Modified Mini-Mental Test.
* Ability to walk independently for at least 6 minutes.
* Receiving physiotherapy and rehabilitation for at least 8 sessions over a 1-month period.
* Having regular access to the internet at home.
* Parent(s) or legal guardian willing to allow the child to participate and able to read and sign the written informed consent form.

Exclusion Criteria:

* Presence of any additional diagnosed neurological disorder other than, or in addition to, Duchenne muscular dystrophy.
* History of any injury and/or surgery within the last 6 months.
* Any cooperation or behavioral problem that prevents completion of the assessment procedures.
* Difficulty in understanding or speaking Turkish.

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Duchenne muscular dystrophy is an X-linked recessive neuromuscular disorder that predominantly affects males. Therefore, only male children with a confirmed diagnosis of DMD are eligible to participate in this study.
Enrollment: 46 (Estimated)
Dates: Start 2026-05-08 (Estimated); Primary Completion 2026-12-21 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) | Baseline, 8 weeks (post-intervention), and 6-month follow-up
  Distance walked in six minutes to assess functional mobility and endurance in ambulatory children w

SECONDARY OUTCOMES:
Modified Upper Extremity Performance Test | Baseline (Day 1), Post-intervention (8 weeks), and 6-month follow-up
  Functional upper extremity performance test quantifying task execution time and efficiency. Higher performance indicates better function.
Repetitive Upper and Lower Extremity Movement Counts | aseline (Day 2), Post-intervention (8 weeks), and 6-month follow-up
  Number of repetitions completed within a standardized time period to assess muscle endurance and functional movement capacity. Higher counts indicate better performance.
Single Breath Counting Test | Baseline (Day 2), Post-intervention (8 weeks), and 6-month follow-up
  Number counted in a single exhalation to assess respiratory function and breath support. Higher values indicate better respiratory capacity.
Pediatric Berg Balance Scale | Baseline (Day 2), Post-intervention (8 weeks), and 6-month follow-up
  Standardized pediatric balance assessment (0-56 range). Higher scores indicate better balance.
Four Square Step Test | Baseline (Day 2), Post-intervention (8 weeks), and 6-month follow-up
  Dynamic balance test measuring time required to sequentially step into four quadrants. Lower times indicate better performance.
ACTIVLIM | Baseline (Day 1), Post-intervention (8 weeks), and 6-month follow-up
  Participation and activity limitation questionnaire assessing perceived difficulty in daily activities. Higher scores reflect lower activity limitation.
Children's Depression Scale | Baseline (Day 2) and Post-intervention (8 weeks)
  Validated pediatric scale assessing depressive symptoms. Higher scores indicate greater depressive symptomatology.
Motivation for Home Exercise (Visual Analog Scale) | Baseline (Day 2) and Post-intervention (8 weeks) and 6 months follow-up
  Motivation rated on a 10 cm visual analog scale. Higher scores reflect higher motivation for home-based exercise participation.
Pediatric Participation Data Collection Tool | Baseline (Day 1) and Post-intervention (8 weeks)
  Structured instrument assessing participation in daily-life activities from pediatric perspective. Higher scores indicate better participation.

IPD SHARING:
Plan to Share IPD: No
Due to pediatric privacy and identifiable rare disease population.